CLINICAL TRIAL: NCT00751829
Title: Comparison of the Efficacy of Olmesartan Medoxomil Versus Nitrendipine on Systolic Blood Pressure in Elderly and Very Elderly Patients With Isolated Systolic Hypertension
Brief Title: Isolated Systolic Hypertension in the Elderly and Very Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Responsible Party: Petra Laeis, Ph.D., Daiichi Sankyo Europe, GmbH
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SE-866/37
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Isolated Systolic Hypertension
MeSH Terms: conditions — Isolated Systolic Hypertension | interventions — Olmesartan Medoxomil; Hydrochlorothiazide; Nitrendipine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): oral olmesartan medoxomil tablets 20 mg or 40 mg once daily for 24 weeks + oral hydrochlorothiazide tablets 12.5 or 25 mg once daily after 12 weeks, if needed to controll BP
  Interventions: Drug: olmesartan medoxomil + hydrochlorothiazide, if necessary
- 2 (Active Comparator): oral nitrendipine tablets 10 or 20 mg taken twice daily for 24 weeks + oral hydrochlorothiazide tablets 12.5 or 25 mg once daily after 12 weeks, if needed to control BP
  Interventions: Drug: nitrendipine + hydrochlorothiazide, if necessary

INTERVENTIONS:
Drug: olmesartan medoxomil + hydrochlorothiazide, if necessary — oral olmesartan medoxomil tablets 20 mg or 40 mg once daily for 24 weeks + oral hydrochlorothiazide tablets 12.5 or 25 mg once daily after 12 weeks, if needed to control BP
  Arms: 1
Drug: nitrendipine + hydrochlorothiazide, if necessary — oral nitrendipine tablets 10 or 20 mg taken twice daily for 24 weeks + oral hydrochlorothiazide tablets 12.5 or 25 mg once daily after 12 weeks, if needed to control BP
  Arms: 2

SUMMARY:
To evaluate the efficacy of long-term treatment of individually optimized doses of olmesartan medoxomil compared to nitrendipine in elderly and very elderly patients with isolated systolic hypertension. The study hypothesis is non-inferiority of olmesartan medoxomil compared to nitrendipine in lowering mean sitting systolic blood pressure after 12 weeks of treatment compared to baseline. The study duration is up to 32 weeks, including a 24-week treatment period. After 12 weeks hydrochlorothiazide may be added to control blood pressure. Efficacy and safety measurements are carried out at up to 15 visits during the trial period.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or older
* Mean sitting BP >160 mmHg and mean sitting dBP<90 mmHg

Exclusion Criteria:

* Secondary hypertension
* Malignant hypertension
* Severe Heart Failure (NYHA III-IV)
* Recent history of myocardial infarction
* Hypersensitivity to study medications
* History of drug or alcohol abuse
* History or evidence of renal disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 417 (Actual)
Dates: Start 2003-07; Primary Completion 2004-10 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Change in mean sitting systolic blood pressure as assessed by conventional BP measurements | 12 weeks

SECONDARY OUTCOMES:
Change in mean sitting systolic blood pressure assessed by conventional BP measurements | After 1, 2, 4, 8, 12, 16, 20, and 24 weeks
Change in mean standing systolic BP, mean sitting diastolic BP and mean standing diastolic BP | after 1, 2, 4, 8, 12, 16, 20, and 24 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter U Witte, MD, Ph.D., Principal Investigator — IMFORM GmbH
Locations (1):
- Munich, Germany